CLINICAL TRIAL: NCT02545010
Title: Phase I Study of Low Dose Whole Abdominal Radiation Therapy (LDWART) in Combination With Weekly Paclitaxel for Platinum Resistant Ovarian Cancer With Predominant Non-visceral Abdominal Disease
Brief Title: Phase I Low Dose WART in Combination With Weekly Paclitaxel for Platinum Resistant Ovarian Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GY01/05/15; 2015/00496 (Other: NHG DSRB)
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LDWART + paclitaxel (Experimental): All patients will receive weekly paclitaxel at a pre specified dose of 80 mg/m2, 70 mg/m2, 60mg/m2 or 50 mg/m2 via intravenous infusion according to institution specific standard practices. Cycles of chemotherapy will be administered weekly without interruption on Days 1,8,15,22,29,36 for a total of 6 weekly cycles in combination with LDWART. LDWART will be given at 60 cGy fractions, twice daily for two days, with a minimum of 4 hours inter fraction interval, starting on day 1 of each cycle of weekly paclitaxel for 6 weeks.
  Interventions: Drug: Paclitaxel; Radiation: LDWART (Low Dose Whole Abdominal Radiation Therapy)

INTERVENTIONS:
Drug: Paclitaxel — All patients will receive weekly paclitaxel at a pre specified dose of 80 mg/m2, 70 mg/m2, 60mg/m2 or 50 mg/m2 via intravenous infusion according to institution specific standard practices.
  Cycles of chemotherapy will be administered weekly without interruption on Days 1,8,15,22,29,36 for a total of 6 weekly cycles in combination with LDWART. Post treatment assessments will be conducted starting Day 43.
  Patients will then continue chemotherapy off trial protocol with weekly paclitaxel without concurrent LDWART starting Day 50 till disease progression, intolerable toxicity, patient refusal or deemed inappropriate to continue treatment by treating physician.
Radiation: LDWART (Low Dose Whole Abdominal Radiation Therapy) — LDWART will be given at 60 cGy fractions, twice daily for two days, with a minimum of 4 hours inter fraction interval, starting on day 1 of each cycle of weekly paclitaxel for 6 weeks.
  LDWART will not be administered if doses of weekly paclitaxel are withheld for any reason since it functions as a "chemosensitizer". LDWART will be administered together weekly paclitaxel immediately at point of recovery from toxicity and patient is deemed to be able to continue with treatment by investigator.

SUMMARY:
Background: Epithelial Ovarian Cancer is the most lethal amongst the gynecologic malignancies and is the fifth leading cause of cancer death in women in the United States.1 Despite initial high response rates, 50% to 75% of women who present with advanced disease suffer relapse and require re treatment2.The optimal treatment for platinum resistant ovarian cancer remains hotly debated. Combination chemotherapy is not favored due to its increased toxicity and lack of convincing benefit when compared to single agent chemotherapy.3,4 Recently, the addition of bevacizumab to single agent chemotherapy in the AURELIA study improved progression free survival (PFS) from 3.4 months to 6.7 months. Response rates were also improved from 11.8% versus 27.3% (p= 0 .001).9 Aim: To determine the maximal tolerated dose (MTD) of weekly paclitaxel in combination with LDWART. The recommended phase II dose (RP2D) will be based on the MTD in this Phase I study. Method: This study is designed as a prospective, single arm phase I study with 3+3 with dose de-escalation and cohort expansion. All patients will receive weekly paclitaxel at a pre specified dose of 80 mg/m2, 70 mg/m2, 60mg/m2 or 50 mg/m2 via intravenous infusion according to institution specific standard practices. Cycles of chemotherapy will be administered weekly without interruption on Days 1,8,15,22,29,36 for a total of 6 weekly cycles in combination with LDWART(Fig.1). LDWART will be given at 60 cGy fractions, twice daily for two days, with a minimum of 4 hours inter fraction interval, starting on day 1 of each cycle of weekly paclitaxel for 6 weeks.(Fig.1). Importance of proposed research: The combination of a LDWART with weekly paclitaxel may improve the efficacy of the current standard weekly paclitaxel in platinum resistant ovarian cancer patients. Potential benefits and risks: The combination may improve treatment response. Adding LDWART may increase treatment risks, but these will be monitored closely.

ELIGIBILITY:
Inclusion Criteria:

* Is capable of understanding the written informed consent, provides signed and witnessed written informed consent, and agrees to comply with protocol requirements.
* Age ≥ 21 years.
* Histologically confirmed and documented epithelial ovarian carcinomas, primary peritoneal carcinomas, or fallopian tube carcinomas.
* Patients must have platinum-resistant disease, (defined as progression within <6 months from completion of a minimum of 4 platinum therapy cycles. The date should be calculated from the last administered dose of platinum therapy).
* Patients must have evidence of measurable intra abdominal disease at point of screening.
* Patients must have disease that is measurable according to RECIST version 1.1 and assessable according to the GCIG CA-125 criteria and require treatment with chemotherapy within 14 days of screening. Target lesions should not be selected in previously irradiated fields unless there is clear evidence of progression
* Performance status of Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2.
* Life expectancy of ≥12 weeks with standard treatment.
* Has adequate organ function at Baseline, including the following (noting that repeated tests at baseline should not be performed unless there are sufficient reasons to assume the patient would meet the inclusion criteria with re-testing):

  1. Absolute neutrophil count ≥1.0 × 109/L
  2. Platelet count ≥100 × 109/L (without transfusions within 21 days prior to Day 1 of Cycle 1)
  3. Hemoglobin ≥9 g/dL
  4. Prothrombin time and partial thromboplastin time within ≤1.5 × upper limit of normal (ULN)
  5. International normalized ratio ≤1.5 × ULN
  6. Total bilirubin ≤1.5 × ULN
  7. Transaminases (aspartate aminotransferase and/or alanine aminotransferase ≤2.5 × ULN (<5 × ULN if liver metastases)
* Has a negative serum pregnancy test 14 days prior to starting study drug plus a negative urine pregnancy test on Day 1, Cycle 1 prior to treatment (applies to females of childbearing potential only).

Exclusion Criteria:

1. General Criteria

   * Is a female patient of childbearing potential, defined as a female physiologically capable of becoming pregnant (including a female whose career, lifestyle, or sexual orientation precludes intercourse with a male partner, and females whose partners have been sterilized by vasectomy or other means), unless they are using a highly effective method for birth control throughout the study and for 12 weeks after the end of treatment. Highly effective methods for birth control include the following:

     1. Total abstinence: This is an acceptable method when this is consistent with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
     2. Female sterilization: The patient has had a surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 6 weeks prior to taking study drug. In case of an oophorectomy alone, the reproductive status of the patient must have been confirmed by follow-up hormone level assessment.
     3. Male partner sterilization: The patient has the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate.

        (For female patients on the study, the vasectomized male partner should be the sole partner for that patient.)

        These patients must also agree to the following:

        Use of a combination of the following (1+2):
        1. Placement of an intrauterine device or intrauterine system
        2. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam, gel, film, or cream, or vaginal suppository Reliable contraception maintained throughout the study and for 12 weeks after study drug discontinuation
     4. Females considered post-menopausal and not of childbearing potential: The definition applies to females who have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone levels >40 mIU/mL (for US only: and estradiol <20 pg/mL) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least 6 weeks prior to starting treatment.

        In the case of oophorectomy alone, only when the reproductive status of the patient has been confirmed by follow-up hormone level assessment is she considered not of childbearing potential.
   * Is a pregnant or nursing (lactating) female, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin laboratory test (>5 mIU/mL). Serum pregnancy test to be assessed within 7 days prior to study treatment start, or within 14 days (with a confirmatory urine pregnancy test within 7 days prior to study treatment start).
   * Is unwilling to or unable to comply with the protocol.
2. Cancer-related

   * Non-epithelial ovarian cancers (Germ cell and stromal ovarian neoplasms)
   * Ovarian tumors with low malignant potential (i.e. borderline tumors).
   * History of other clinically active malignancy within 5 years of enrollment, except for tumors with a negligible risk for metastasis or death, such as adequately controlled basal-cell carcinoma or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix or breast.
   * Has central nervous system metastasis, unless previously treated with surgery, whole-brain radiation or stereotactic radiosurgery, and stable disease for at least 8 weeks without steroid use for at least 4 weeks prior to the first dose of weekly paclitaxel.
   * Symptomatic intestinal obstruction requiring surgical intervention or bowel rest.
3. Prior, current or planned treatment:

   * Previous treatment with 3 or more anticancer regimens.
   * Has used other investigational drugs within 4 weeks or five half-lives (whichever is longer) prior to the first dose of study treatment.
   * Has received prior radiation therapy within 4 weeks, or limited field radiation within 2 weeks, prior to starting study drug, or the side effects of such therapy have not resolved to ≤Grade 1.
   * Has had a major surgical procedure within 4 weeks from starting the study drug. Patient has not fully recovered from all surgery-related complications to ≤Grade 1
4. Prior or concomitant conditions or procedures:

   * History or evidence upon physical / neurological examination of CNS disease unrelated to cancer, unless adequately treated with standard medical therapy (e.g. uncontrolled seizures).
   * Pre-existing peripheral neuropathy ≥ CTC grade.
   * Serious active infection requiring intravenous antibiotics and/or hospitalization at study entry.
   * Known grade 3 or ≥ hypersensitivity to any of the study drugs or excipients.
   * Evidence of any other medical conditions (such as psychiatric illness, etc.), physical examination or laboratory findings that may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment-related complications.
   * Has a history of interstitial lung disease, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, or pulmonary hypersensitivity pneumonitis.
   * Has severe or unstable medical conditions such as heart failure, ischemic heart disease, uncontrolled hypertension, uncontrolled diabetes mellitus, psychiatric condition, an ongoing cardiac arrhythmia requiring medication (≥Grade 2, according to National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] Version 4.03), or any other significant or unstable concurrent medical illness that in the opinion of the investigator would preclude protocol therapy.
   * Has a known history of human immunodeficiency virus seropositivity or other active bacterial, viral, or fungal infections. Hep B or C positive patients on anti-viral treatment are eligible for the study

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerated dose (MTD) of weekly paclitaxel in combination with LDWART | Up to 6 weeks from initiation of treatment
  The maximum tolerated dose (MTD) of weekly paclitaxel and LDWART is defined as the lowest dose cohort of weekly paclitaxel and LDWART where ≥ 2 out of initial 3 or ≥ 2 out of total 6 patients in any cohort develops a DLT

SECONDARY OUTCOMES:
Objective response rate (ORR) | From the time of their first treatment with weekly paclitaxel and LDWART till 30 days from end of last treatment
  Objective Response Rate will be assessed with RECIST v1.1 and GCIG CA-125 response criteria.
Progression Free Survival (PFS) | From the time of their first treatment with weekly paclitaxel and LDWART till 1 year from end of last treatmen
  Progression Free Survival will be calculated from the date of initiation of therapy to the first day when the RECIST (version 1.1) criteria for progressive disease (PD) are met.
Dose limiting toxicity (DLT) | From the time of their first treatment with weekly paclitaxel and LDWART till 30 days from end of last treatment
  Dose-limiting toxicities (DLT) occurring in the first 3 weeks of treatment in the phase I dose-escalation stage will be used in dose de-escalation decisions. Safety and toxicity will be assessed in all patients using the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 to determine the MTD and RP2D.

CONTACTS AND LOCATIONS:
Overall Officials: David SP Tan, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Pujade-Lauraine E, Hilpert F, Weber B, Reuss A, Poveda A, Kristensen G, Sorio R, Vergote I, Witteveen P, Bamias A, Pereira D, Wimberger P, Oaknin A, Mirza MR, Follana P, Bollag D, Ray-Coquard I. Bevacizumab combined with chemotherapy for platinum-resistant recurrent ovarian cancer: The AURELIA open-label randomized phase III trial. J Clin Oncol. 2014 May 1;32(13):1302-8. doi: 10.1200/JCO.2013.51.4489. Epub 2014 Mar 17. PMID 24637997
- [Background] Kunos CA, Sill MW, Buekers TE, Walker JL, Schilder JM, Yamada SD, Waggoner SE, Mohiuddin M, Fracasso PM. Low-dose abdominal radiation as a docetaxel chemosensitizer for recurrent epithelial ovarian cancer: a phase I study of the Gynecologic Oncology Group. Gynecol Oncol. 2011 Feb;120(2):224-8. doi: 10.1016/j.ygyno.2010.10.018. PMID 21075438
- [Derived] Ngoi NYL, Heong V, Tang JI, Choo BA, Kumarakulasinghe NB, Lim D, Low M, Lim SE, Lim YW, Leong YH, Tseng M, Tong PSY, Ilancheran A, Low JJH, Ng J, Thian YL, Koh V, Tan DSP. Phase 1 Study of Low-Dose Fractionated Whole Abdominal Radiation Therapy in Combination With Weekly Paclitaxel for Platinum-Resistant Ovarian Cancer (GCGS-01). Int J Radiat Oncol Biol Phys. 2021 Mar 1;109(3):701-711. doi: 10.1016/j.ijrobp.2020.09.059. Epub 2020 Oct 9. PMID 33045316